CLINICAL TRIAL: NCT05112900
Title: SCALE-UP Counts: A Health Information Technology Approach to Increasing COVID-19 Testing in Elementary and Middle Schools Serving Disadvantaged Communities
Brief Title: Health Information Technology for COVID-19 Testing in Schools (SCALE-UP Counts)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Yelena Wu, Associate Professor, Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB_00143340; 1OT2HD108097-01 (NIH)
Record Dates: First submitted 2021-11-01; First posted 2021-11-09 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
Keywords: Adolescents; Behavioral Research; Screening
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A Parallel study using short time frames (<1 month) and iterative evaluation cycles. The proposed trial will compare the efficacy of text messaging (TM) and text messaging plus health navigation (TM+HN) versus usual care. All randomizations will take place on the individual level at the beginning of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Participants will only receive unidirectional public service announcement-type text messaging on COVID-19 testing every 3 weeks such as recommendation to obtain COVID-19 testing if exposed, experience symptoms, or have an interest in preemptive testing and information on testing options through the school or district.
- Text Messaging (TM) (Experimental): This arm consists of a text message (TM) prompt asking if a participant has COVID-19 symptoms or if a participant has been exposed to a person who has tested positive for COVID-19. If a participant responds yes, they will receive a TM prompt for immediate testing and to re-test. Participants will also be asked if they have an interest in preemptive testing, regardless of symptoms or exposure Participants will be provided with information on testing options. After 24 hours, the participant will receive another TM that asks if they tested and what their results are. After 3 days, participants will be prompted to re-test.
  Interventions: Behavioral: Text Messaging (TM)
- Text Messaging plus Health Navigation (TM+HN) (Experimental): TM+HN consists of the same intervention as TM with the addition of health navigation services based on non-compliance. Participants will be evaluated as non-compliant if they had reported symptoms, contact, or interest in testing and then stop responding to text messages or respond that they did not test. Health navigator (HN) calls will be conducted using Motivation and Problem Solving (MAPS).
  Interventions: Behavioral: Text Messaging + Health Navigation (TM+HN)

INTERVENTIONS:
Behavioral: Text Messaging (TM) — [see arm/group descriptions]
  Arms: Text Messaging (TM)
Behavioral: Text Messaging + Health Navigation (TM+HN) — [see arm/group descriptions]
  Arms: Text Messaging plus Health Navigation (TM+HN)

SUMMARY:
This project will address key testing challenges in Utah schools by building on collaborations with public school districts, private schools, charter schools and with Utah Department of Health on coronavirus disease (COVID-19) testing and existing infrastructure. The study team will work closely with schools and the Utah public health system to implement and test a shovel-ready and scalable health information technology approach that delivers automated text messages (TM) to students' parents around COVID-19 testing. In addition, some parents will receive a health navigator (HN) follow-up to ensure that tests are completed. Families will be offered the recently FDA-approved in-home serial testing approach if accessing in-person testing is a challenge. While this project is focused on COVID-19 testing, in the case that the COVID-19 vaccination becomes more relevant or is the priority of the school, the study team is able to tailor the intervention to focus on the vaccine as well. The outcomes in this study utilized parent/student reported data. Staff data were also collected but will not be reflected in primary outcome analyses.

DETAILED DESCRIPTION:
Intervention: Randomization of parent/student participants will take place upon enrollment in the study. Participants are assigned to either usual care (UC), text messaging (TM), or text messaging plus health navigation (TM+HN).

Participants included are those who did not opt-out of the study. Participants eligible for Randomization will either be assigned to 1) Usual Care (control, approximately 20% of participants), 2) Text Message (TM, approximately 40% of participants), or 3) Text Message plus Health Navigation (TM+HN, approximately 40% of participants).

Usual Care participants will only receive unidirectional and fixed public service announcement-type text messaging on COVID-19 testing every 3 weeks (e.g., recommendation to obtain COVID-19 testing if exposed or experience symptoms; information on testing options through the school or district).

TM consists of a more intensive, bidirectional text message prompt asking if a participant has COVID-19 symptoms or if a participant has been exposed to a person that has tested positive for COVID-19, or if the participant has interest in preemptive testing. If a participant responds yes, they will receive a TM prompt for immediate testing and to re-test. Participants will be provided with information on testing options for COVID-19. After 24 hours, the participant will be asked if they tested and what their results are. After 3 days, participants will be prompted to re-test. If a participant had interest in preemptive testing, they will be asked if testing was completed after 7 days. Testing and re-testing prompts will be adjusted through the study to mirror public health guidance on testing strategies.

TM+HN consists of the same intervention as TM with the addition of health navigation services based on participant non-compliance. Participants will be evaluated as non-compliant if they had reported symptoms, contact, or interest in testing and then stop responding to text messages or respond that they did not test. Health navigator (HN) calls will be conducted using Motivation and Problem Solving (MAPS). MAPS is an empirically validated proactive coaching approach used to address barriers and motivate participants to utilize testing options if they are experiencing COVID-19 symptoms, have been exposed to someone that has tested positive for COVID-19, or reported interest in preemptive testing.

Assessments: The study team will collect survey data from parents at pre- and post-intervention as well as throughout the trial. COVID-19 test results of participants will be collected through self-report as well as through results reported to the "Ellume" testing app. Additionally, the study team will conduct stakeholder interviews with students, parents, and staff on ways to improve the interventions to better meet their needs and preferences.

Addendum to study allocation ratio: Change of allocation for participants eligible for Randomization

• The study's allocation ratio was changed on 7/20/22. The original allocation ratio for the study was 20% usual care with the remaining 80% randomly assigned equally to the TM and TM+HN groups. The new allocation ratio was 50% randomly assigned to control with the remaining 50% randomly assigned equally to the TM and TM+HN groups. The reason for the change in allocation ratio is that the study team observed low numbers of participants reporting any COVID-19 testing. Thus, in order to optimize statistical power to be able to compare the control group to both experimental groups (TM and TM+HN) together in end-of-study analyses, the allocation ratio was changed. For schools that were enrolled in the study prior to this allocation ratio change, individuals in that school who had already been assigned a study condition maintained their original assignment. To account for this change in allocation, we will adjust for the allocation ratio for when the participant was randomized, within the model.

Addendum to outcome measures timeline: Change of survey timeline of outcomes for eligible participants

• The survey distribution timeline was changed 9/27/22. The 6-month survey was not distributed (due to an electronic distribution error) and the timing of this survey was changed to 9 months post intervention enrollment. Additionally, the 1-month survey was only distributed in Year 1 of the study. Newly enrolled participants in Year 2 (as of 8/1/22) did not receive the 1-month survey. The purpose of the 1-month survey was to complete an early assessment of the intervention to determine if any changes were needed based on participant feedback, and thus was not needed in the second year of the study. Enrolled participants that did not complete the baseline survey were sent a follow up survey at the end of the study to collect demographic and other outcomes data. A final survey distributed at the end of the study was also added in order to assess accessibility, feasibility, and other outcomes.

ELIGIBILITY:
Inclusion Criteria:

Students

* Attends school at any of the participating schools from the districts the research team is working with

Parents

* Legal guardian/parent of the student
* Has a functioning cellular phone that can receive calls and text messages

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7122 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Wu, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Wu YP, Chipman JJ, Kolp L, Stump TK, Kuzmenko TV, Del Fiol G, Haaland B, Kaphingst KA, Brooks R, Hersh AL, Brady HL, Lundberg KJ, Wan N, Carroll C, Orleans B, Wirth J, Wetter DW. Mobile Intervention for Increasing COVID-19 Testing in K-12 Schools Serving Disadvantaged Communities: Randomized Controlled Trial of SCALE-UP Counts. J Med Internet Res. 2025 Nov 11;27:e79775. doi: 10.2196/79775. PMID 41217804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Utah K-12 schools were recruited between October 2021 and March 2023. Recruitment focused on Title 1 schools and schools in underserved communities. Parents were eligible to participate if they had a functioning cell phone that could receive/send text messages. This study used an opt-out design. Schools provided parent telephone numbers who were contacted by text with an initial opportunity to opt-out. Those who did not opt out within 24 hours of the initial message were automatically enrolled.
Pre-assignment Details: 1. Randomization Error- Multiple records per phone number, randomized more than once
  2. Excluded for other reasons- No home address, Opt-out before randomization
Groups:
- Usual Care: Participants will only receive unidirectional, static, public service announcement-type text messaging on COVID-19 testing every 3 weeks such as recommendation to obtain COVID-19 testing if exposed, experience symptoms, or have an interest in preemptive testing and information on testing options through the school or district. Participants were informed on how to access test kits through the participating school and were provided with an email address to request test kits by direct mail from the study team.
- Text Messaging (TM): This arm consists of a text message (TM) prompt asking if a participant has COVID-19 symptoms or if a participant has been exposed to a person who has tested positive for COVID-19. If a participant responds yes, they will receive a TM prompt for immediate testing and to re-test. Participants will also be asked if they have an interest in preemptive testing, regardless of symptoms or exposure Participants will be provided with information on testing options. After 24 hours, the participant will receive another TM that asks if they tested and what their results are. After 3 days, participants will be prompted to re-test.
  Participants were informed on how to access test kits by pick up from the participating school and provided an email address to request test kits by direct mail from the study team through text messaging.
- Text Messaging and Health Navigation (TM+HN): This arm consists of the same text message prompts as the TM group with the addition of health navigator services (TM+HN) through a brief telephone call. These calls will be conducted using Motivation and Problem Solving (MAPS). Participants in this arm that interacted with the text messaging system by indicating an interest in testing but did not report test completion were deemed "non-responders". Non-responders in this group received the phone call from a health navigator to assess testing barriers.
  Participants were informed on how to access test kits by pick up from the participating school and provided an email address to request test kits by direct mail from the study team through text messaging.
Period: Overall Study
Arm/Group | Usual Care | Text Messaging (TM) | Text Messaging and Health Navigation (TM+HN)
Started | 2588 | 2270 | 2264
Completed | 1628 | 1349 | 1296
Not Completed | 960 | 921 | 968
Not completed — Withdrawal by Subject | 960 | 921 | 968

BASELINE CHARACTERISTICS:
Population: Characteristics provided are at the individual student level. Students did not receive text messages or participate directly. Parent reported data was provided at the household-level. Parents were eligible to participate on the condition they had a student enrolled. Characteristics are provided at the student level to capture the student population the study served and accounts for the higher number of participants than reported in Participant Flow and randomization.
Groups:
- Text Messaging + Health Navigation (TM+HN): This arm consists of the same text message prompts as the TM group with the addition of health navigator services (TM+HN) through a brief telephone call. These calls will be conducted using Motivation and Problem Solving (MAPS). Participants in this arm that interacted with the text messaging system by indicating an interest in testing but did not report test completion were deemed "non-responders". Non-responders in this group received the phone call from a health navigator to assess testing barriers.
  Participants were informed on how to access test kits by pick up from the participating school and provided an email address to request test kits by direct mail from the study team through text messaging.
- Total: Total of all reporting groups
Arm/Group | Usual Care | Text Messaging (TM) | Text Messaging + Health Navigation (TM+HN) | Total
Number analyzed (Participants) | 2367 | 2187 | 2166 | 6720
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2367 | 2187 | 2166 | 6720
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 1166 | 1092 | 1066 | 3324
  Sex/Gender: Male | 1197 | 1092 | 1099 | 3388
  Sex/Gender: Unknown | 4 | 3 | 1 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian/NA | 17 | 29 | 30 | 76
  Race/Ethnicity: Asian | 108 | 128 | 124 | 360
  Race/Ethnicity: Native Hawaiian or Pacific Islander | 69 | 77 | 66 | 212
  Race/Ethnicity: Black or African American | 89 | 85 | 71 | 245
  Race/Ethnicity: White | 1329 | 1277 | 1316 | 3922
  Race/Ethnicity: Hispanic or Latino | 752 | 589 | 558 | 1899
  Race/Ethnicity: Unknown or Not Reported | 3 | 2 | 1 | 6
Free/Reduced Lunch of students [Number; unit: percent] — Percent of students who qualify for free or reduced lunch
  percent | 51.70 | 52.86 | 52.20 | 52.25

OUTCOME MEASURES:

1. Primary Outcome: Testing Uptake- The Number of Valid Responses That Confirmed COVID-19 Testing Was Completed by Households
Description: The study team will examine whether students and/or members of their household tested by analyzing the number of valid responses that confirmed COVID-19 testing was completed by households
Time Frame: Monthly (up to 16-months post-baseline)
Population: Unique participants that responded to text messages on COVID-19 testing completion.
Measure: Mean (Standard Deviation); unit: Valid response to message on testing
Groups:
- Text Messaging Plus Health Navigation: This arm consists of the same text message prompts as the TM group with the addition of health navigator services (TM+HN) through a brief telephone call. These calls will be conducted using Motivation and Problem Solving (MAPS). Participants in this arm that interacted with the text messaging system by indicating an interest in testing but did not report test completion were deemed "non-responders". Non-responders in this group received the phone call from a health navigator to assess testing barriers.
  Participants were informed on how to access test kits by pick up from the participating school and provided an email address to request test kits by direct mail from the study team through text messaging.
Arm/Group | Usual Care | Text Messaging (TM) | Text Messaging Plus Health Navigation
Number analyzed (Participants) | 966 | 789 | 770
Valid response to message on testing | .1603 (.3669) | .2552 (.4361) | .2484 (.4322)

2. Secondary Outcome: Missed School Days
Description: The study team will examine the number of missed school days enrolled students missed due to COVID-19 related reasons (e.g., exposure, testing).
Time Frame: Monthly (up to 16-months post-baseline)
Population: The population analyzed are participants that responded to the surveys assessing for missed school days. Not all participants responded to this survey.
Measure: Mean (Standard Deviation); unit: Number of missed school days
Arm/Group | Usual Care | Text Messaging (TM) | Text Messaging Plus Health Navigation
Number analyzed (Participants) | 797 | 803 | 968
Number of missed school days | .25 (1.11) | .37 (1.27) | .38 (1.17)

ADVERSE EVENTS:
Time Frame: 16 months
Description: This study was a text message based study that had little risk to participants. There are zero series adverse events, all-cause mortality, or other adverse events to report.
Arm/Group | Usual Care | Text Messaging (TM) | Text Messaging + Health Navigation (TM+HN)
All-Cause Mortality (participants affected / at risk) | 0/2367 | 0/2187 | 0/2166
Serious Adverse Events (participants affected / at risk) | 0/2367 | 0/2187 | 0/2166
Other Adverse Events (participants affected / at risk) | 0/2367 | 0/2187 | 0/2166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT05112900/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT05112900/SAP_001.pdf